CLINICAL TRIAL: NCT02422758
Title: Prewarming Effect in Preventing Perioperative Hypothermia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cibele Cristina Tramontini Fuganti, Cibele Cristina Tramontini Fuganti, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 38320814.2.0000.5393
Record Dates: First submitted 2015-04-08; First posted 2015-04-21 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Hypothermia
Keywords: hypothermia; perioperative nursing; prewarming; prevention and control
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Prewarming 3M™ BairHugger™Blanket (Experimental): Patients will have the whole body covered with the3M™ Bair Hugger™ Preoperative & Outpatient Care Blanket of forced air warming system for 20 minutes, at average power.Tympanic temperature will be measured, through electronic infrared tympanic thermometer GENIUS 2. Patients will be warmed with 3M™ Bair Hugger™ Upper Body Blanket, during intraoperative period.
  Interventions: Device: 3M™ Bair Hugger™ Preoperative & Outpatient Care Blanket
- Passive Prewarming (Placebo Comparator): Passive prewarming with a cotton sheet and blanket for 20 minutes. Tympanic temperature will be measured, through electronic infrared tympanic thermometer GENIUS 2. Patients will be warmed with 3M™ Bair Hugger™ Upper Body Blanket, during intraoperative period.
  Interventions: Other: Passive Prewarming

INTERVENTIONS:
Device: 3M™ Bair Hugger™ Preoperative & Outpatient Care Blanket — 3M™ Bair Hugger™Preoperative & Outpatient Care Blanket will cover the whole body. Patients will be prewarmed for 20 minutes with forced air warming system. Unit will be at average power.
  Other Names: 3M™ Bair Hugger™Blanket Model 110
  Arms: Active Prewarming 3M™ BairHugger™Blanket
Other: Passive Prewarming
  Arms: Passive Prewarming

SUMMARY:
Perioperative hypothermia brings numerous and recognized postoperative complications. Active warming intraoperatively helps to maintain body temperature in the postoperative period, but there are few studies in Brazil, assessing the effect of prewarming in maintaining normothermia. It is believed that prewarming with forced air warming system keep the body temperature during intra and post-operative. This study aims to evaluate the effect on prewarming maintaining body temperature of patients undergoing elective surgery of Gynecology specialty using the forced air warming system. The study is experimental design, controlled type randomized clinical trial, with simple blinding for patients. Eighty adult patients undergoing gynecological surgery in the art, with a surgical time of at least an hour will be randomized and allocated into experimental groups - prewarming system with forced air warming system for 20 minutes, and control - Prewarming with sheet and blanket for 20 minutes. The patients will be kept warm during the anesthetic-surgical procedure. The measurement of temperature will be using a tympanic thermometer. Participants will be followed from receiving the surgical center to the end of surgery. Data will be recorded in validated instrument. Data analysis will be used the Model Linear Mixed Effects and the Structure Error Auto-Regressive.

DETAILED DESCRIPTION:
Maintaining the patient in the perioperative normothermia is a challenge for surgical and nursing staff. Despite advances in the development of new technologies for the prevention of perioperative hypothermia, this event still happens in the operating room of the health services To prevent patient's body temperature loss, passive and active cutaneous warming methods can be used. Passive methods prevent loss of body heat through the heat transfer block, as blankets, clothes and cotton sheets; however, there is evidence to show that although assist in maintaining body temperature, passive methods alone are not effective.

Active warming methods are effective in keeping the perioperative normothermia. Among the different technologies available we emphasize the circulating water mattress, the forced air warming system and the carbon fiber resistive heating blankets.

Based on these and due to the lack of research in the Brazilian reality on effective measures for the prevention of perioperative hypothermia, among these, prewarming, and the finding guided by the professional experience that just directed investment for the maintenance of body temperature patient in the perioperative period, in health services, justified the conduct of this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years;
* Undergoing elective surgery with duration of at least one hour in the gynecological specialty with open technique;
* Under general, regional or combined anesthesia.

Exclusion Criteria:

* Patients with a body temperature above or below 36oC 37,5oC at the reception of the operating room.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of prewarming in maintaining body temperature of patients undergoing elective gynecologic surgery. | intraoperative
  The temperature will be evaluated throughout the operation and maintenance will be verified at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cibele Cristina T Fuganti, RN, MS, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Background] Andrzejowski J, Hoyle J, Eapen G, Turnbull D. Effect of prewarming on post-induction core temperature and the incidence of inadvertent perioperative hypothermia in patients undergoing general anaesthesia. Br J Anaesth. 2008 Nov;101(5):627-31. doi: 10.1093/bja/aen272. Epub 2008 Sep 26. PMID 18820248
- [Background] ASSOCIATION OF PERIOPERATIVE REGISTERED NURSES (AORN). Recommended practices for the prevention of unplanned perioperative hypothermia. In: ASSOCIATION OF PERIOPERATIVE REGISTERED NURSES. Perioperative standards and recommended practices. Denver (USA): Association of periOpertive Registered Nurses; 2009.p. 491-504.
- [Background] De Witte JL, Demeyer C, Vandemaele E. Resistive-heating or forced-air warming for the prevention of redistribution hypothermia. Anesth Analg. 2010 Mar 1;110(3):829-33. doi: 10.1213/ANE.0b013e3181cb3ebf. Epub 2009 Dec 30. PMID 20042439
- [Background] Fettes S, Mulvaine M, Van Doren E. Effect of preoperative forced-air warming on postoperative temperature and postanesthesia care unit length of stay. AORN J. 2013 Mar;97(3):323-8. doi: 10.1016/j.aorn.2012.12.011. PMID 23452697
- [Background] Galvao CM, Marck PB, Sawada NO, Clark AM. A systematic review of the effectiveness of cutaneous warming systems to prevent hypothermia. J Clin Nurs. 2009 Mar;18(5):627-36. doi: 10.1111/j.1365-2702.2008.02668.x. PMID 19239533
- [Background] Leslie K, Sessler DI. Perioperative hypothermia in the high-risk surgical patient. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):485-98. doi: 10.1016/s1521-6896(03)00049-1. PMID 14661653
- [Background] Tramontini CC, Graziano KU. Hypothermia control in elderly surgical patients in the intraoperative period: evaluation of two nursing interventions. Rev Lat Am Enfermagem. 2007 Jul-Aug;15(4):626-31. doi: 10.1590/s0104-11692007000400016. PMID 17923980
- [Background] Weirich TL. Hypothermia/warming protocols: why are they not widely used in the OR? AORN J. 2008 Feb;87(2):333-44. doi: 10.1016/j.aorn.2007.08.021. PMID 18262000
- [Background] NATIONAL INSTITUTE FOR HEALTH AND CLINICAL EXCELLENCE (NICE). Clinical practice guideline - The management of inadvertent perioperative hypothermia in adults. 2008, 567p.
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665
- [Background] Wartzek T, Muhlsteff J, Imhoff M. Temperature measurement. Biomed Tech (Berl). 2011 Oct;56(5):241-57. doi: 10.1515/BMT.2011.108. PMID 21988157
- [Background] Knaepel A. Inadvertent perioperative hypothermia: a literature review. J Perioper Pract. 2012 Mar;22(3):86-90. doi: 10.1177/175045891202200302. PMID 22493869
- [Background] Wagner D, Byrne M, Kolcaba K. Effects of comfort warming on preoperative patients. AORN J. 2006 Sep;84(3):427-48. doi: 10.1016/s0001-2092(06)63920-3. PMID 17004666
- [Background] Lynch S, Dixon J, Leary D. Reducing the risk of unplanned perioperative hypothermia. AORN J. 2010 Nov;92(5):553-62; quiz 563-5. doi: 10.1016/j.aorn.2010.06.015. PMID 21040819
- [Background] Poveda Vde B, Galvao CM. [Hypothermia in the intraoperative period: can it be avoided?]. Rev Esc Enferm USP. 2011 Apr;45(2):411-7. doi: 10.1590/s0080-62342011000200016. Portuguese. PMID 21655792
- [Background] Galvao CM, Liang Y, Clark AM. Effectiveness of cutaneous warming systems on temperature control: meta-analysis. J Adv Nurs. 2010 Jun;66(6):1196-206. doi: 10.1111/j.1365-2648.2010.05312.x. PMID 20546353
- [Background] Esnaola NF, Cole DJ. Perioperative normothermia during major surgery: is it important? Adv Surg. 2011;45:249-63. doi: 10.1016/j.yasu.2011.03.007. PMID 21954692
- [Background] POVEDA, V. B.; MARTINEZ, E. Z.; GALVÃO, C. M. Métodos ativos de aquecimento para a prevenção de hipotermia no período intraoperatório: revisão sistemática. Rev. Latino-Am. Enfermagem, v.20, n.1, p. 183-191, 2012.
- [Background] de Brito Poveda V, Clark AM, Galvao CM. A systematic review on the effectiveness of prewarming to prevent perioperative hypothermia. J Clin Nurs. 2013 Apr;22(7-8):906-18. doi: 10.1111/j.1365-2702.2012.04287.x. Epub 2012 Sep 17. PMID 22978458
- [Derived] Fuganti CCT, Martinez EZ, Galvao CM. Effect of preheating on the maintenance of body temperature in surgical patients: a randomized clinical trial. Rev Lat Am Enfermagem. 2018 Oct 25;26:e3057. doi: 10.1590/1518-8345.2559.3057. PMID 30379244